CLINICAL TRIAL: NCT02397603
Title: Peri-neural Dexmedetomidine as an Adjuvant to Bupivacaine-induced Paravertebral Block in Patients Undergoing Thoracotomy
Brief Title: Peri-neural Dexmedetomidine as an Adjuvant to Bupivacaine Induced Paravertebral Block in Patients Undergonig Thoracotomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Professor Mohamed Abdulatif Mohamed, Professor of Anesthesiology & Surgical Intensive Care, Faculity of Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N-16-2015
Record Dates: First submitted 2015-03-15; First posted 2015-03-25 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Acute Post-thoracotomy Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bupivacaine saline group (Active Comparator): This group of patients will receive 20 ml bupivacaine plus 0.5 ml normal saline perineurally in the paravertebral catheter
  Interventions: Drug: Bupivacaine saline
- Dexmedetomidine- bupivacaine group (Active Comparator): This group of patients will receive 20 ml bupivacaine plus 0.5 ml (50 microgram) dexmedetomidine administered perineurally in the paravertebral catheter.
  Interventions: Drug: dexmedetomidine bupivacaine

INTERVENTIONS:
Drug: dexmedetomidine bupivacaine — perineural dexmedetomidine as an adjuvant to bupivacaine induced thoracic paravertebral block
  Arms: Dexmedetomidine- bupivacaine group
Drug: Bupivacaine saline — perineural bupivacaine saline mixture in the thoracic paravertebral catheter
  Arms: bupivacaine saline group

SUMMARY:
This study evaluates the effect of adding dexmedetomidine as an adjuvant to bupivacaine in patients undergoing thoracotomy when administered peri-neurally in thoracic paravertebral space.

DETAILED DESCRIPTION:
Thoracotomy is associated with severe postoperative pain that could be reduced with an aggressive analgesic therapy in the early postoperative period. The use of thoracic paravertebral block is an effective analgesic approach for post-thoracotomy pain. Several local anesthetic adjuvants have been reported to extend the duration of paravertebral block.

Alpha-2 agonists including dexmedetomidine appear to be the most effective in this context. The study will include an intervention group which will receive a combination of 20 ml bupivacaine 0.5% and dexmedetomidine 0.5 ml (50 microgram). The control group will receive 20 ml bupivacaine 0.5% plus 0.5 ml normal saline perineurally. Thoracic paravertebral catheter will be inserted preoperatively. Visual analogue pain score will be assessed at different intervals.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists physical status class ||or |||.
* Patients scheduled for elective thoracotomy.

Exclusion Criteria:

* Pneumonectomy, decortication, pleural biopsy.
* Additional chest wall resection.
* Emergency surgery.
* Central and peripheral neuropathies.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Duration of first loading preoperative dose of paravertebral injectate | One day
  Time interval between initiation of the paravertebral block and the time to first rescue analgesia

SECONDARY OUTCOMES:
Duration of surgery and anesthesia | Intraoperative period, up to 3-4 hours
  Times from start of anesthesia and surgery to the conclusion of surgical intervention
End tidal isoflurane | Duration of anesthesia, up to 3-4 hours
  Average End-tidal isoflurane concentration required to maintain stable hemodynamics
Total intraoperative fentanyl requirements | Intraoperative period, up to 3-4 hours
  The total dose of fentanyl required during the surgical procedure to maintain hemodynamic stability
Total intraoperative ephedrine and atropine requirements | Intraoperative period, up to 3-4 hours
  The total amounts of ephidrine and atropine required for the treatment of possible reduction of arterial blood pressure or heart rate
Total intraoperative crystalloid requirements | Intraoperative period, up to 3-4 hours
  The total volume of intraoperative fluids in ml required to maintain hemodynamic stability
Recovery time | Immediate postoperative period, up to 2 hour
  the time interval between discontinuation of isoflurane and the patient first response to verbal commands
Pain intensities at rest and during coughing as assessed by 0-10 VAS score | Over 48 hours postoperatively
  Pain scores will be assessed using the 11-points visual analogue pain score (VAS) where 0 indicates no pain and 10 indicates the worst pain.
Total doses of bupivacaine, dexmedetomidine, and morphine | 48 hours postoperatively
  The total doses of three medications will be recorded and compared in the intervention and control groups
Number of paravertebral to-up injections | 48 hours postoperatively
  The number of to-up doses of bupivacaine required to maintain adequate postoperative analgesia over 48 hours postoperatively
Side effects | 48 hours postoperatively
  Patients will be monitored for the possible reductions in arterial blood pressure and heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdulatif, MD., Principal Investigator — Professor of anesthesia, surgical intensive care and pain management cairo university
Locations (1):
- Kasr Alainy Hospital Cairo University, Giza, Egypt

REFERENCES:
- [Result] Marhofer D, Kettner SC, Marhofer P, Pils S, Weber M, Zeitlinger M. Dexmedetomidine as an adjuvant to ropivacaine prolongs peripheral nerve block: a volunteer study. Br J Anaesth. 2013 Mar;110(3):438-42. doi: 10.1093/bja/aes400. Epub 2012 Nov 15. PMID 23161360